CLINICAL TRIAL: NCT02648230
Title: PrEssure wiRe Compared to Microcatheter-based Sensing Technology For the Evaluation of cORonary Fractional Flow Reserve Measurements
Brief Title: PrEssure wiRe Compared to Microcatheter-based Sensing Technology For the Evaluation of FFR Measurements
Acronym: PERFORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Ajay Kirtane, Associate Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAQ1712
Record Dates: First submitted 2015-12-23; First posted 2016-01-06 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Ischemia; Angina
Keywords: Ischemia; Fractional Flow Reserve; Stent
MeSH Terms: conditions — Ischemia; Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pressure wire and Microcatheter (Experimental): All subjects enrolled will have both an FFR done measured by a pressure wire (PW) and then again by a microcatheter (MC).
  Interventions: Device: St. Jude Medical Pressure Wire; Device: ACIST Navvus Microcatheter

INTERVENTIONS:
Device: St. Jude Medical Pressure Wire — FFR measurement will be obtained with a PW with the FFR measurement obtained by using a MC within the same subject across the same target lesion at the same time
  Other Names: PW
Device: ACIST Navvus Microcatheter — FFR measurement will be obtained with a MC with the FFR measurement obtained by using a PW within the same subject across the same target lesion at the same time
  Other Names: MC

SUMMARY:
The model by which physicians measure the lack of blood flow in the vessels that supply blood to the heart muscle is called Fractional Flow Reserve (FFR). FFR is the measurement of the pressure across the vessels that supply blood to the heart. These are known as the coronary arteries. This study involves comparing two FFR wires, the St. Jude Medical Pressure Wire (PW) and the ACIST Navvus Microcatheter (MC) to check the accuracy of the devices. FFR allows real-time estimation of the effects of a narrowed vessel, whereas standard angiography can underestimate or overestimate narrowing, because it only visualizes contrast (the different areas of color) inside a vessel.

DETAILED DESCRIPTION:
Fractional flow reserve (FFR) measurement by pressure wire (PW) under hyperemic conditions has become the invasive gold standard for determining the physiologic extent of cardiac ischemia, and which has been validated in several clinical outcomes studies as a way of optimizing case selection for percutaneous coronary intervention (PCI). More recently a microcatheter (MC)-based sensor measurement of fractional flow reserve has been introduced. Small scale in-vivo comparisons have been performed suggesting the utility of this approach to measure FFR,but these data are limited and have not been independently validated. This non-randomized, prospective study is designed to evaluate the accuracy of MC-based FFR measurement to the PW standard in lesions subjected to FFR assessment in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patient provides signed written informed consent before any study-specific procedure.
3. Undergoing coronary angiography, for silent ischemia, stable angina, acute coronary syndrome, or other acceptable indication per the local standard of care.
4. Angiographically significant (>50% visual estimation) stenosis present in at least one native coronary artery.
5. Undergoing FFR assessment for standard clinical or diagnostic indications

Exclusion Criteria:

1. Aorto-ostial lesion location within 3 mm of the aorta junction (both right and left).
2. Vessel(s) and lesion(s) not amenable for PCI, for example diffuse disease.
3. Currently participating in another clinical study that interferes with study results.
4. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure.
5. Any other medical condition that in the opinion of the investigator will interfere with patient safety or study results.
6. High degree A-V block, sinus node disease.
7. Known hypersensitivity to adenosine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12-08 (Actual); Study Completion 2016-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Kirtane, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled between December 2015 to December 2016.
Groups:
- Pressure Wire and Microcatheter: All subjects enrolled will have both a fractional flow reserve (FFR) done measured by a pressure wire (PW) and then again by a microcatheter (MC).
  St. Jude Medical Pressure Wire: FFR measurement will be obtained with a PW with the FFR measurement obtained by using a MC within the same subject across the same target lesion at the same time
  ACIST Navvus Microcatheter: FFR measurement will be obtained with a MC with the FFR measurement obtained by using a PW within the same subject across the same target lesion at the same time
Period: Overall Study
Arm/Group | Pressure Wire and Microcatheter
Started | 74
Completed | 74
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pressure Wire and Microcatheter
Number analyzed (Participants) | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 38
  More than one race | 0
  Unknown or Not Reported | 27

OUTCOME MEASURES:

1. Primary Outcome: Mean Fractional Flow Reserve (FFR)
Description: The mean FFR will be measured with the pressure catheter (PC) to be compared against the mean FFR measured with a standard Pressure Wire (PW) within the same subject across the same target lesion at the same time. Fractional flow reserve measurement involves determining the ratio between the maximum achievable blood flow in a diseased coronary artery and the theoretical maximum flow in a normal coronary artery.
Time Frame: Through study completion (an average of an hour)
Measure: Mean (Inter-Quartile Range); unit: ratio
Arm/Group | Pressure Wire and Microcatheter
Number analyzed (Participants) | 74
ratio
  Pressure Wire | 0.84 [0.78 to 0.89]
  Pressure Catheter (microcatheter) | 0.79 [0.73 to 0.85]

ADVERSE EVENTS:
Arm/Group | Pressure Wire and Microcatheter
All-Cause Mortality (participants affected / at risk) | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74
Other Adverse Events (participants affected / at risk) | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes